CLINICAL TRIAL: NCT03764111
Title: Ultrasound Image Quality Comparison Between an Inexpensive Handheld Ultrasound Machine and a Large Mobile Ultrasound System
Brief Title: Comparing an Inexpensive Handheld Ultrasound Machine and a Large Mobile Ultrasound System
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000024151
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- large mobile ultrasound system: the ultrasound transducer is based on piezoelectric technology.
  Interventions: Device: Large Mobile Ultrasound System
- handheld ultrasound machine: The handheld device utilizes Capacitive micro-machined ultrasound transducers (CMUTs) instead of piezoelectric technology
  Interventions: Device: Handheld Ultrasound Machine

INTERVENTIONS:
Device: Large Mobile Ultrasound System — 30 spine images, 15 Transverse abdominis muscle and 30 Obstetric images (i.e placenta, uterine blood flow, etc) images will be obtained using the large mobile ultrasound system.
  Other Names: Sonosite - M turbo
  Groups: large mobile ultrasound system
Device: Handheld Ultrasound Machine — 30 spine images, 15 Transverse abdominis muscle and 30 Obstetric images (i.e placenta, uterine blood flow, etc) images will be obtained using the handheld device.
  Other Names: Butterfly iQ device
  Groups: handheld ultrasound machine

SUMMARY:
To assess the quality of images and diagnostic ability of a handheld device under two thousand dollars against those of a bigger and more expensive ultrasound machine.

DETAILED DESCRIPTION:
Ultrasound technology is frequently used to obtain information, usually at patients bedside. The images obtained are used to guide procedure (i.e central line placement, epidural needle guidance) or to make diagnosis (i.e abnormal placentation, presence of pneumothorax). Given that the majority of this procedures and diagnosis are made at bedside, the ideal ultrasound machine should be portable, lightweight, and within an acceptable price range. Our current ultrasound machine (Sonosite - M turbo) has a price range from 15,000-20,000 dollars, not including the different probes that are needed to obtain images at different depths in the human body. Much of the cost is due to the ultrasound transducers, which have been traditionally based on piezoelectric technology. Such probes work by passing current through a piezoelectric crystal (typically quartz) that then vibrates rapidly and generates an ultrasound pulse. Creating crystal arrays is difficult and often requires hand-manufacturing. Furthermore, this technology is analog and requires downstream analog-to-digital processing hardware. Together, these characteristics increase device costs and restrict the broader dissemination of ultrasound technology.

Recently, the Butterfly iQ company created an ultrasound that is portable and at a price of slightly under two thousand dollars it allows the physician to obtain images for diagnostic and/or procedural guidance using a single probe. The company was able to significantly reduced the cost and the need for additional probes by utilizing Capacitive micro-machined ultrasound transducers (CMUTs). Essentially instead of relying on the use of specific piezoelectric crystals (current ultrasound technology), they are using a micro-chip technology to emit the vibrations that would be used to form an image. Butterfly Network has developed a CMUT imaging device that has been designed to be compliant with all applicable FDA safety regulations (see section II.C), while enabling increased portability and real-time smartphone-based image review due to the integrated circuit design. The Butterfly device was FDA-approved as of October 2017. The proposed study will compare the images acquired by the Butterfly iQ and our current Sonosite M-turbo US.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing a routine obstetric scan or requesting a transverse abdominis block, labor epidural or spinal for cesarean delivery.

Exclusion Criteria:

* Body Mass Index (BMI) > 45

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients between the ages of 18 and 45 presenting for cesarean delivery requesting a transverse abdominis block, epidural, or in need of an obstetric US.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Ultrasound image quality-resolution | Prior to start of active labor or before elective cesarean delivery
  Images will be rated on a 10-point Likert-type scale; higher scores indicate better image quality.
Ultrasound image quality-details | Prior to start of active labor or before elective cesarean delivery
  Images will be rated on a 10-point Likert-type scale; higher scores indicate better image quality.
Ultrasound image quality-total image quality | Prior to start of active labor or before elective cesarean delivery
  Images will be rated on a 10-point Likert-type scale; higher scores indicate better image quality.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gonzalez, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khuri-Yakub BT, Oralkan O. Capacitive micromachined ultrasonic transducers for medical imaging and therapy. J Micromech Microeng. 2011 May;21(5):54004-54014. doi: 10.1088/0960-1317/21/5/054004. PMID 21860542